CLINICAL TRIAL: NCT04856839
Title: Phenotypes, Biomarkers and Pathophysiology in Syringomyelia
Brief Title: Clinical Outcome in Patients With Syringomyelia（COPSM）
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Fengzeng Jian, director of neurospine department, Xuanwu hospital, Xuanwu Hospital, Beijing
Other Study IDs: XWCOPSM
Record Dates: First submitted 2021-04-17; First posted 2021-04-23 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Syringomyelia/Hydromyelia
Keywords: Syringomyelia, Biomarker，Electrophysiology
MeSH Terms: conditions — Syringomyelia | interventions — Electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, cerebral spinal fluid, saliva, urine, biopsy and autopsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- syringomyelia group
  Interventions: Diagnostic Test: high throughput sequencing and electromyography
- Other neurodegenerative diseases: such as hydrocephalus
  Interventions: Diagnostic Test: high throughput sequencing and electromyography
- Normal group
  Interventions: Diagnostic Test: high throughput sequencing and electromyography

INTERVENTIONS:
Diagnostic Test: high throughput sequencing and electromyography — Whole Genome Sequencing, Whole Exome Sequencing, Transcriptomics, Proteomics, Metabolomics

SUMMARY:
The aim of this study is to determine the clinical spectrum and natural progression of Syringomyelia (SM) and related disorders in a prospective single center study, identify digital, imaging and molecular biomarkers that can assist in diagnosis and therapy development and study the etiology and molecular mechanisms of these diseases.

DETAILED DESCRIPTION:
Syringomyelia is a chronic central spinal cord injury, which is characterized by dilation of the central canal of the spinal cord. At present, the treatment of syringomyelia is mainly through surgical decompression to restore the disturbance of cerebrospinal fluid circulation. Due to the heterogeneity of the etiology of syringomyelia, almost all published studies on the clinical outcome and prognostic factors of syringomyelia are relatively limited, and most of them are retrospective. It is not clear which is the most reliable predictor of clinical outcome. Therefore, the researchers conducted this prospective cohort study to identify the occurrence, development and outcome of syringomyelia and determine the main prognostic factors through clinical scales, biomarkers and electrophysiology.

At study visits a standardized clinical examination will be performed including application of clinical rating scales. At all study visits, patients will be asked to donate biosamples; biomaterial collection is optional and participants can elect to participate in sampling of blood, urine, CSF, and/or a muscle biopsy.

Optionally, additional examinations may be performed including imaging, neurophysiological examination, analysis of patient or observer reported outcomes and analysis to characterize molecular biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* patients who was diagnosed as syringomyelia including: Chiari malformation， Basilar Impression， subarachnoid obstruction， patient not received surgical or interventional treatment before， patient willing and able to participate in the registry，
* Hydrocephalus or other neurodegenerative disease and normal subjects.

Exclusion Criteria:

* patient received surgical treatment or interventional treatment before
* patient is pregnant
* patient unable to complete follow-up
* patient with other spinal lesions
* other nervous system diseases

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients who was diagnosed as syringomyelia including: Chiari malformation、Basilar Impression、subarachnoid obstruction
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change of the spinal cord function | 1 day before operation and 3 days, 3 months, 12 months postoperation
  American Spinal Injury Association(ASIA) Score for evaluating the spinal cord function

SECONDARY OUTCOMES:
molecular profiling results | 1 day before operation and 3 days, 3 months postoperation
  Change From Baseline in molecular at postoperation
Electrophysiology results | 1 day before operation and 3 days, 3 months postoperation
  included：electromyography and evoked potential; Change From Baseline in Electrophysiology at postoperation
the rates of syrinx reduction | 3 days, 3 months postoperation
  defined as a reduction of the syrinx diameter or length in MRI
Chicago Chiari outcome scale (CCOS) | 3 days, 3 months, 12 months postoperation
  Pain symptoms,Nonpain symptoms,Functionality,Complications, 4-16, higher scores mean a better outcome.
Visual Analog Scale (VAS) | 1 day before operation and 3 days, 3 months, 12 months postoperation
  degree of the pain, 1-10, higher scores mean a worse outcome
Klekamp and Sammi syringomyelia scale | 1 day before operation and 3 days, 3 months, 12 months postoperation
  for evaluating the spinal cord function, higher scores mean a better outcome
modified Japanese Orthopaedic Association Scores (mJOA) | 1 day before operation and 3 days, 3 months, 12 months postoperation
  Motor function， sensory， bladder function；for evaluating the spinal cord function；0-17， higher scores mean a better outcome
Incidence of perioperative complications | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Fengzeng Jian, M.D., Study Director — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] CreveCoeur TS, Yahanda AT, Maher CO, Johnson GW, Ackerman LL, Adelson PD, Ahmed R, Albert GW, Aldana PR, Alden TD, Anderson RCE, Baird L, Bauer DF, Bierbrauer KS, Brockmeyer DL, Chern JJ, Couture DE, Daniels DJ, Dauser RC, Durham SR, Ellenbogen RG, Eskandari R, Fuchs HE, George TM, Grant GA, Graupman PC, Greene S, Greenfield JP, Gross NL, Guillaume DJ, Haller G, Hankinson TC, Heuer GG, Iantosca M, Iskandar BJ, Jackson EM, Jea AH, Johnston JM, Keating RF, Kelly MP, Khan N, Krieger MD, Leonard JR, Mangano FT, Mapstone TB, McComb JG, Menezes AH, Muhlbauer M, Oakes WJ, Olavarria G, O'Neill BR, Park TS, Ragheb J, Selden NR, Shah MN, Shannon C, Shimony JS, Smith J, Smyth MD, Stone SSD, Strahle JM, Tamber MS, Torner JC, Tuite GF, Wait SD, Wellons JC, Whitehead WE, Limbrick DD. Occipital-Cervical Fusion and Ventral Decompression in the Surgical Management of Chiari-1 Malformation and Syringomyelia: Analysis of Data From the Park-Reeves Syringomyelia Research Consortium. Neurosurgery. 2021 Jan 13;88(2):332-341. doi: 10.1093/neuros/nyaa460. PMID 33313928
- [Background] Nakajima M, Rauramaa T, Makinen PM, Hiltunen M, Herukka SK, Kokki M, Musialowicz T, Jyrkkanen HK, Danner N, Junkkari A, Koivisto AM, Jaaskelainen JE, Miyajima M, Ogino I, Furuta A, Akiba C, Kawamura K, Kamohara C, Sugano H, Tange Y, Karagiozov K, Leinonen V, Arai H. Protein tyrosine phosphatase receptor type Q in cerebrospinal fluid reflects ependymal cell dysfunction and is a potential biomarker for adult chronic hydrocephalus. Eur J Neurol. 2021 Feb;28(2):389-400. doi: 10.1111/ene.14575. Epub 2020 Nov 1. PMID 33035386
- [Background] Klekamp J. Surgical treatment of Chiari I malformation--analysis of intraoperative findings, complications, and outcome for 371 foramen magnum decompressions. Neurosurgery. 2012 Aug;71(2):365-80; discussion 380. doi: 10.1227/NEU.0b013e31825c3426. PMID 22569058
- [Background] Roser F, Ebner FH, Liebsch M, Dietz K, Tatagiba M. A new concept in the electrophysiological evaluation of syringomyelia. J Neurosurg Spine. 2008 Jun;8(6):517-23. doi: 10.3171/SPI/2008/8/6/517. PMID 18518671
- [Background] Sadler B, Wilborn J, Antunes L, Kuensting T, Hale AT, Gannon SR, McCall K, Cruchaga C, Harms M, Voisin N, Reymond A, Cappuccio G, Brunetti-Pierri N, Tartaglia M, Niceta M, Leoni C, Zampino G, Ashley-Koch A, Urbizu A, Garrett ME, Soldano K, Macaya A, Conrad D, Strahle J, Dobbs MB, Turner TN, Shannon CN, Brockmeyer D, Limbrick DD, Gurnett CA, Haller G. Rare and de novo coding variants in chromodomain genes in Chiari I malformation. Am J Hum Genet. 2021 Mar 4;108(3):530-531. doi: 10.1016/j.ajhg.2021.01.014. No abstract available. PMID 33667397
- [Background] Guan J, Yuan C, Zhang C, Ma L, Yao Q, Cheng L, Liu Z, Wang K, Duan W, Wang X, Wang Z, Wu H, Chen Z, Jian F. A novel classification and its clinical significance in Chiari I malformation with syringomyelia based on high-resolution MRI. Eur Spine J. 2021 Jun;30(6):1623-1634. doi: 10.1007/s00586-021-06746-y. Epub 2021 Feb 5. PMID 33544223